CLINICAL TRIAL: NCT05777395
Title: Comparison of Maitland Oscillatory Mobilizations With Kaltenborn Sustained Stretch Mobilizations in Cervicogenic Headache Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/1
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive conventional physical therapy along with Maitland oscillatory mobilizations and the second will receive Kaltenborn sustained stretch mobilizations with conventional physical therapy. Both groups will be recruited concurrently.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not be aware of which group the participant belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maitland + Conventional PT Group (Experimental): Participants of this group will receive the conventional physical therapy protocol mentioned above. In addition to this, they will receive Maitland oscillatory mobilizations. 3 sets of 15 repetitions. Each set is of 30 seconds and each repetition is given in 2 seconds.
  * Frequency: 3 times a week for 2 weeks. 6 sessions in total.
  * Mobilizations will be performed in Grade 1 initially and then progressed to Grade 2 and 3.
  * Techniques used are postero-anterior unilateral vertebral pressure and Maitland rotation.
  Interventions: Procedure: Maitland Oscillatory Mobilization; Procedure: Conventional therapy
- Kaltenborn + Conventional PT Group (Experimental): Participants of this Group will receive the conventional physical therapy protocol mentioned above. In addition to this, they will receive Kaltenborn sustained stretch mobilizations. 3 sets of 15 repetitions for 3 seconds.
  * Frequency: 3 times a week for 2 weeks. 6 sessions in total.
  * Mobilizations will be performed in Grade 1 and then progressed to 2 and 3.
  * Kaltenborn technique used will be atlas-axis rotation.
  Interventions: Procedure: Kaltenborn Sustained Stretch Mobilization; Procedure: Conventional therapy

INTERVENTIONS:
Procedure: Maitland Oscillatory Mobilization — Maitland Posteroanterior unilateral vertebral pressure and Maitland cervical rotation technique will be used.3 sets of 15 repetitions. Each set is of 30 seconds and each repetition is given for 2 seconds.
  Arms: Maitland + Conventional PT Group
Procedure: Kaltenborn Sustained Stretch Mobilization — Kaltenborn sustained stretch mobilizations. 3 sets of 15 repetitions for 3 seconds.
  * Frequency: 3 times a week for 2 weeks. 6 sessions in total.
  * Mobilizations will be performed in Grade 1 and then progressed to 2 and 3.
  * Kaltenborn technique used will be atlas-axis rotation
  Arms: Kaltenborn + Conventional PT Group
Procedure: Conventional therapy — Moist heat, TENS, Neck Muscle Stretching, Neck muscle isometrics

SUMMARY:
Cervicogenic headache is a common headache that causes disability and affects everyday activities. Headache related disorders are the second most common reason for years lived with disability all over the world. According to the latest International Headache Society model, cervicogenicheadache (CGH) is a secondary headache having C1-C2 dysfunction. There is marked limitation in cervical ROM specially rotation. Treatment indicated involves use of electrotherapy and thermal modalities. In addition, use of different manual therapy techniques are advocated to eliminate the root cause i.e. C1-C2 dysfunction. Maitland mobilizations for cervical spine have been found to be effective in treating CGH patients. Maitland mobilizations uses oscillatory mobilizations and has four grades. Kaltenborn, on the other hand, applies sustained stretches and has 3 grades.So, the study will be focusing on comparing the effectiveness of these two mobilizations on cervicogenic headache patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Both males and females
* Unilateral headache with no shift of side
* C1-C2 dysfunction
* Headache with neck stiffness
* Headache at least once a month in the last 3 months
* Positive flexion rotation test (Rotation restriction is greater than 10 degrees)
* Headache with a score of at least 4 in the Numeric pain rating scale

Exclusion Criteria:

* Cervical spondylosis
* Headache of non-cervical origin
* Dizziness or visual disturbance
* Cervical radiculopathy/ nerve root involvement/ disc herniation
* Cervical instability/ fracture
* Vertebrobasilar insufficiency
* Thoracic outlet syndrome
* Cervical spine surgery
* Cervical spondylolisthesis
* Spinal infection or tumors
* Osteoporosis
* History of trauma
* Metabolic disorders
* Rheumatoid Arthritis
* Inflammatory Arthritis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  Pain will be measured on the basis of Numeric Pain Rating Scale score.
Cervical range of motion | 2 weeks
  Cervical rotation will be measured through CROM device

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan